CLINICAL TRIAL: NCT05027126
Title: Comparison of Bioavailability of Dexketoprofen-Vit B vs Dexketoprofen (Stadium®), Dose 25 mg in Healthy Subjects, of Both Genders, Under Fasting Conditions
Brief Title: Comparison of Bioavailability of Dexketoprofen-Vit B vs Dexketoprofen, in Healthy Subjects, Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DEXK-Sil No. 101-18
Record Dates: First submitted 2021-08-25; First posted 2021-08-30 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Healthy
Keywords: Dexketoprofen; Trometamol; Cyanocobalamin; Thiamine; Pyridoxine; Pharmacokinetic; Bioavailability; Fixed-dose combination (FDC); Bioequivalence
MeSH Terms: interventions — dexketoprofen trometamol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Dexketoprofen (Stadium®) (Active Comparator): Reference Drug Pharmaceutical Form: Tablets Dosage: 25 mg Administration way: oral
  Interventions: Drug: Dexketoprofen 25 MG
- Group B: Fixed dose Dexketoprofen-Vitamin B Complex (Experimental): Fixed dose combination: Pharmaceutical Form: capsule Dosage: 25 mg of Dexketoprofen + Cyanocobalamin, Thiamine,and Pyridoxine. Administration way: oral
  Interventions: Drug: Fixed dose Dexketoprofen-Vitamin B Complex

INTERVENTIONS:
Drug: Dexketoprofen 25 MG — Pharmaceutical Form: Tablets Dosage: 25 mg Adminstration way: Oral
  Other Names: (Stadium®)
  Arms: Group A: Dexketoprofen (Stadium®)
Drug: Fixed dose Dexketoprofen-Vitamin B Complex — Pharmaceutical Form: capsule Dosage: 25 mg of Dexketoprofen + Cyanocobalamin 500 µg, Thiamine 100 mg, Pyridoxine 50 mg. Administration way: oral
  Other Names: DEXK / VITB
  Arms: Group B: Fixed dose Dexketoprofen-Vitamin B Complex

SUMMARY:
Bioavailability comparison study with a cross-over desing, 2x2, open, prospective and longitudinal, at a single dose with two treatments, two periods, two sequences with an elimination (washout) period of 7 days and a number of 36 healthy subjects, of both genders, under fasting conditions, of reference tablets of Dexketoprofen 25 mg (Stadium®), elaborated by Grimann, S.A. de C.V., and capsule test drug with Dexketoprofen 25 mg- Vitamin B complex elaborated by Laboratorios Silanes S.A. de C.V.

DETAILED DESCRIPTION:
The study was designed to recruit 36 healthy subjects considering a 2x2 design, where each subject received both treatments and was its own control. The time was adjusted considering the half-life of the drugs to be evaluated. Healthy subjects of both genders were selected since no relevant pharmacokinetic differences related to gender had been reported for the study drug. The aim of the study was to comparatively evaluate, in the same individuals the plasma concentrations of Dexketoprofen 25 mg from two pharmaceutical formulations; reference tablets of Dexketoprofen 25 mg ( Stadium®), elaborated by Grimann, S.A. de C.V., and capsule test drug with Dexketoprofen 25 mg- Vitamin B complex elaborated by Laboratorios Silanes S.A. de C.V.

ELIGIBILITY:
Inclusion Criteria:

* That the patient gives informed consent in writing.
* Be accepted by the COFEPRIS research subjects registry base.
* Subjects without subordination relationship with the researchers or sponsor. - Subjects of both genders, aged between 18 and 55, Mexican.
* No history of hypersensitivity or related drug allergies.
* Body mass index between 18 and 27 kg / m2
* Healthy subjects, according to the results of the complete clinical history, electrocardiogram and the integration of the results of the clinical analyzes, carried out in certified clinical laboratories, without alterations that, at the discretion of the Principal Investigator, require medical intervention as a consequence.
* Subjects with negative results for immunological tests (Anti-HIV (Human immunodeficiency virus), Anti-hepatitis B and C, VDRL (venereal disease reaction level)).
* Subjects with negative results in qualitative tests for the detection of drugs of abuse: tetrahydro-cannabinoids, cocaine and
* Research subject that presents alterations in the vital signs recorded during the selection.amphetamines.
* Negative (qualitative) pregnancy test in the case of women of childbearing age without bilateral tubal obstruction or hysterectomy.
* In the case of women of childbearing age, the subject must sign a letter of commitment not to pregnancy and have a birth control method, including barrier methods, non-hormonal intrauterine device or bilateral tubal obstruction.

Exclusion Criteria:

* Subjects with a recent history (3 months) or evidence on physical examination of gastrointestinal, renal, hepatic, endocrine, respiratory, cardiovascular, dermatological or hematological disease that could affect the pharmacokinetic study of the investigational product.
* Subjects who have been exposed to drugs known as liver enzyme inducers or inhibitors or who have taken potentially toxic drugs within 30 days prior to the start of the study.
* Subjects who have received any medication for 7 days prior to the start of the study.
* Subjects who have been hospitalized for any problem during the three months prior to the start of the study.
* Subjects who have been rejected for their registration in the COFEPRIS research subject registry database, for having participated in a clinical study within the three months prior to the start of the study.
* Subjects who have received investigational drugs within 60 days prior to the study.
* Subjects allergic to the drug under study or related drugs.
* Subjects who have ingested alcohol or beverages containing xanthines (coffee, tea, cocoa, chocolate, cola soft drinks) or who have ingested charcoal-grilled foods or grapefruit or cranberry juice, at least 10 hours before the start of the study or who have smoked tobacco within 24 hours prior to the start of the internment period.
* Subjects who have donated or lost 450 mL or more of blood within the 60 days prior to the start of the study.
* Subjects with a history of drug and / or alcohol abuse according to the DSM-IV-TR ( Diagnostic and Statistical Manual of Mental Disorders) Criteria.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration following the treatment (Cmax) | Baseline, 0.16, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 14.00 and 24.00 hours
  Evaluate the fixed dose pharmacokinetics profile of Dexketoprofen-Vitamin B, employing the maximum observed concentration following the treatment (Cmax).
The area under the curve from time zero to the last measurable concentration (AUC 0-t) | Baseline, 0.16, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 14.00 and 24.00 hours
  Evaluate the fixed dose pharmacokinetics profile of Dexketoprofen-Vitamin B, employing the area under the curve from time zero to the last measurable concentration (AUC 0-t)using the linear trapezoidal method.
The area under the curve from time zero to infinity calculated (AUC 0-inf) | Baseline, 0.16, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 14.00 and 24.00 hours
  Evaluate the fixed dose pharmacokinetics profile of Dexketoprofen-Vitamin B, employing the area under the curve from time zero to infinity (AUC 0-inf), estimated by adding the quotient of the last concentration measured between ke.
Time of the maximum measured concentration (Tmax). | Baseline, 0.16, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 14.00 and 24.00 hours
  Evaluate the fixed dose pharmacokinetics profile of Dexketoprofen-Vitamin B, employing time of the maximum measured concentration (Tmax)
Elimination rate (Ke) | Baseline, 0.16, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 14.00 and 24.00 hours
  Evaluate the fixed dose pharmacokinetics profile of Dexketoprofen-Vitamin B, employing the elimination rate (Ke), calculated by log-linear regression of the final phase of elimination
Elimination half-life (t 1/2) | Baseline, 0.16, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 14.00 and 24.00 hours
  Evaluate the fixed dose pharmacokinetics profile of Dexketoprofen-Vitamin B, employing the elimination half-life (t 1/2) by dividing 0.693 / ke.

SECONDARY OUTCOMES:
The frequency of adverse events | 2 days
  The percentage of frequency of appearance of each adverse event was evaluated.
Adverse events | 2 days
  Any adverse event were classified by severity, treatment and its relationship with the study drug was evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes Garza Ocaña, M.D, Principal Investigator — Department of Pharmacology and Toxicology of the Faculty of Medicine of the U.A.N.L; Eduardo J Tamez de la O, M.D, Principal Investigator — Department of Pharmacology and Toxicology of the Faculty of Medicine of the U.A.N.L
Locations (1):
- Laboratorio Silanes, S.A. de C.V., Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barbanoj MJ, Gich I, Artigas R, Tost D, Moros C, Antonijoan RM, Garcia ML, Mauleon D. Pharmacokinetics of Dexketoprofen Trometamol in Healthy Volunteers After Single and Repeated Oral Doses. J Clin Pharmacol. 1998 Dec;38(S1):33S-40S. doi: 10.1002/jcph.1998.38.s1.33. PMID 29023869
- [Background] Barbanoj MJ, Antonijoan RM, Gich I. Clinical pharmacokinetics of dexketoprofen. Clin Pharmacokinet. 2001;40(4):245-62. doi: 10.2165/00003088-200140040-00002. PMID 11368291
- [Background] Schuirmann DJ. A comparison of the two one-sided tests procedure and the power approach for assessing the equivalence of average bioavailability. J Pharmacokinet Biopharm. 1987 Dec;15(6):657-80. doi: 10.1007/BF01068419. PMID 3450848
- See also: Spanish Agency for Medicines and Health Products (AEMPS). Ministry of Health, Social Policy and Equality. Technical sheet Metamizole ratiopharm 575 mg hard capsules — https://cima.aemps.es/cima/dochtml/ft/72769/FT_72769.html
- See also: STADIUM. Drugs. — https://www.medicamentosplm.com/Home/productos/stadium_tabletas/160/101/9884/210
- See also: Official Mexican standard that establishes the tests and procedures to demonstrate that a drug is interchangeable. Requirements to which the Authorized Third Parties that carry out the interchangeability tests must be subject. — http://www.dof.gob.mx/nota_detalle.php?codigo=5314833&fecha=20/09/2013
- See also: R Core Team (2019). R: A language and environment for statistical computing. — http://www.r-project.org/